CLINICAL TRIAL: NCT03227692
Title: Randomized Controlled Study Comparing iASSIST Knee System Versus Conventional Instrumentation
Brief Title: Persona TKA With iASSIST Knee System and iASSIST Knee System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: K.CR.I.AP.16.39
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Results first posted 2020-03-19 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: At surgery, intervention group using iASSIST Knee system. At surgery, conventional group not using iASSIST Knee system.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Persona TKA with iASSIST Knee system (Investigational group) or Persona TKA with conventional instrumentation (Control group). The randomization scheme is based on equal numbers per group. The randomization will occur via a random number generator (computer) using blocked randomization procedure. The PI or his/her team does not have influence on the randomization scheme. Sealed opaque envelopes, which will be prepared based on predetermined randomization assignment, will be provided to each study site before study initiation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Persona with iASSIST Knee (Experimental): Having total knee arthroplasty (Persona Knee System) surgery with the use of a navigation system iASSIST Knee.
  Interventions: Device: Persona Knee System; Procedure: Total Knee Arthroplasty; Device: iAssist Knee
- Persona without iASSIST Knee (Active Comparator): Having total knee arthroplasty surgery (Persona Knee System) with the use of conventional surgical instruments, and without a navigation system iASSIST Knee.
  Interventions: Device: Persona Knee System; Procedure: Total Knee Arthroplasty

INTERVENTIONS:
Device: Persona Knee System — Osteoarthritis will be enrolled and randomly assigned into one of two treatment groups. Patients in investigational group will be treated with total knee arthroplasty and the accelerometer-based navigational device. Patients in control group will be treated with total knee arthroplasty with conventional instrumentation.
  Other Names: Persona Knee
Procedure: Total Knee Arthroplasty — Damaged cartilage due to degerative arthritis is replaced by knee joint prosthesis.
  Other Names: TKA
Device: iAssist Knee — Osteotomy of TKA is navigated by iAssist system, iAssist requires pin inserted in bone.
  Arms: Persona with iASSIST Knee

SUMMARY:
The purpose of this study is to compare the accuracy of knee component alignment between patients operated with iASSIST Knee (Investigational group) versus patients operated without iASSIST Knee (Control group) using the same implant system.

DETAILED DESCRIPTION:
Objective： To compare the accuracy of knee component alignment between patients operated with iASSIST Knee (Investigational group) versus patients operated without iASSIST Knee (Control group) using the same implant system.

Endpoint： Primary： The alignment accuracy of the knee femoral and tibial components at 6 months for the investigational group compared to the control group.

Secondary：Health Status after TKA, Operating Room efficiency and Complication rate after TKA for the investigational group compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a patient must meet all of the following criteria.

* Knee (either unilateral or bilateral) osteoarthritis (varus deformity only)
* Male or female
* At least 20 years of age
* Patients willing to return for follow-up evaluations.

Study Specific Requirements for Principal Investigator/Site

* Principal Investigator (PI) must have experience of at least 5 TKAs of iASSIST Knee with Persona and Persona conventional instrument system before any study specific activities.
* Site has sufficient resources to take limb CT scanning at 6 months follow-up visit.

Exclusion Criteria:

Absolute contraindications include:

* Knee degenerative diseases other than knee osteoarthritis (such as necrosis/rheumatoid arthritis)
* Too severe OA deformation (FTA: > 190 degrees/< 175 degrees)
* Active infection (or within 6 weeks after infection)
* Sepsis
* Osteomyelitis
* Any type of implant is inserted in the affected side of lower extremity
* Hip and/or foot disease on the affected side

Additional contraindications include:

* Uncooperative patient or patient with neurologic disorders who are incapable of following directions
* Diagnosed osteoporosis or osteomalacia
* Metabolic disorders which may impair bone formation
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy or neuromuscular disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toshihiro Ohdera, M.D., Principal Investigator — Fukuoka Orthopaedic Hospital
Locations (3):
- Japan (3):
  - Sumitomo Hopital, Osaka, Osaka
  - Japanese Red Cross Medical Center, Shibuya City, Tokyo
  - Yamaguchi Prefectural Grand Medical Center, Hōfu, Yamaguchi

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Persona With iASSIST Knee | Persona Without iASSIST Knee
Started | 47 | 46
Completed | 42 | 41
Not Completed | 5 | 5
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 4 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Persona With iASSIST Knee | Persona Without iASSIST Knee | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (9.0) | 76.1 (9.0) | 74.8 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 31 | 66
  Male | 7 | 10 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 42 | 41 | 83
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 42 | 41 | 83
KSS - Objective Score [Mean (Standard Deviation); unit: score on scale] — KSS-Objective score is physician-derived component and allows for more than 100 points in patients with greater than 125° of flexion and a stable painless knee as outlined below. Lowest possible score is 0.
  Higher score means better outcomes.
  score on scale | 34.8 (20.2) | 36.1 (19.8) | 35.4 (19.9)
KSS-Patient Satisfaction [Mean (Standard Deviation); unit: score on a scale] — KSS-Patient Satisfaction is patient-derived score and is a five-question 40-point scale that is collected preoperatively and at each follow-up visit. Lowest possible score is 0.
  Higher score means better outcomes.
  score on a scale | 12.7 (6.3) | 15.1 (6.1) | 13.9 (6.3)
KSS-Function Score [Mean (Standard Deviation); unit: score on a scale] — KSS-function score is patient-derived score and composed of four subgroups and has a maximum score of 100.
  "Walking and Standing" has a maximum value of 30 points, "Standard Activities" has a maximum of 30 points, "Advanced Activities" has a maximum of 25 points and "Discretionary Activities" has a maximum of 15 points.
  Lowest possible score is 0. Higher score means better outcomes.
  score on a scale | 38.5 (0.2) | 39.1 (17.6) | 38.8 (18.9)
KSS-Patient Expectation [Mean (Standard Deviation); unit: score on scale] — KSS-Patient Expectations is patient-derived score and is a three-question fifteen-point scale that is collected pre-operatively and post-operatively. The pre-operative questions reflect the patient's opinion on the extent to which the patient expects that operation will improve knee pain, and ability to perform activities of daily living and recreational activities. The post-operative questions reflect the extent to which postoperative outcome has met the patient's pre-operative expectations with respect to pain and function.
  The score ranges from 3 to 15. Higher score means better outcomes.
  score on scale | 13.1 (2.0) | 12.9 (1.7) | 13.0 (1.9)
Oxford Knee Score [Mean (Standard Deviation); unit: score on scale] — Patient Reported Outcome specific for knee disease. Score range from 0 to 48. Higher score means better outcome.
  score on scale | 22.0 (9.1) | 25.0 (8.4) | 23.5 (8.8)
EQ-5D-3L [Mean (Standard Deviation); unit: score on a scale] — EQ-5D is patient reported outcome measure to score patient's health related quality of life with minimum score of -0.111 and maximum score of 1.000.
  Higher score means better outcomes.
  score on a scale | 0.6 (0.2) | 0.6 (0.1) | 0.6 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Alignment Accuracy of the Knee Femoral Components in Coronal Plain
Description: Ratio of subject, whose knee implant is positioned within 3 degrees from perpendicular to mechanical axis of lower extremity, is compared between groups by CT data taken at 6 month after surgery.
Time Frame: Postoperative 6 months
Population: Patients who have CT data at 6 month after surgery were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Persona With iASSIST Knee | Persona Without iASSIST Knee
Number analyzed (Participants) | 42 | 41
Participants
  within 3 degrees | 39 | 36
  outlier | 3 | 5

2. Primary Outcome: Number of Participants With Alignment Accuracy of the Knee Femoral Components in Sagittal Plain
Description: as for outcome 1
Time Frame: Postoperative 6 months
Population: Patients who have CT data at 6 month after surgery were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Persona With iASSIST Knee | Persona Without iASSIST Knee
Number analyzed (Participants) | 42 | 41
Participants
  within 3 degrees | 36 | 24
  outlier | 6 | 17

3. Primary Outcome: Number of Participants With Alignment Accuracy of the Knee Tibial Components in Coronal Plain
Description: as for outcome 1
Time Frame: Postoperative 6 months
Population: Patients who have CT data at 6 month after surgery were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Persona With iASSIST Knee | Persona Without iASSIST Knee
Number analyzed (Participants) | 42 | 41
Participants
  within 3 degrees | 32 | 23
  outlier | 10 | 18

4. Primary Outcome: Number of Participants With Alignment Accuracy of the Knee Tibial Components in Sagittal Plain
Description: Ratio of subject, whose knee implant is positioned within 3 degrees from preoperatively determined target angle, is compared between groups by CT data taken at 6 month after surgery.
Time Frame: Postoperative 6 months
Population: Patients who have CT data at 6 month after surgery were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Persona With iASSIST Knee | Persona Without iASSIST Knee
Number analyzed (Participants) | 42 | 41
Participants
  within 3 degrees | 34 | 32
  outlier | 8 | 9

5. Secondary Outcome: Surgery Time
Description: Surgery time from skin incision to closure
Time Frame: Intraoperative, an average of 2 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Persona With iASSIST Knee | Persona Without iASSIST Knee
Number analyzed (Participants) | 47 | 46
minutes | 125.1 (34.6) | 114.2 (32.4)

6. Secondary Outcome: Number of Instrument Trays Used
Description: Number of instrument trays used instraoperatively. This number includes number of Total Knee Arthroplasty specific instrument tray, does not include other general surgical instruments/kits.
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: trays
Arm/Group | Persona With iASSIST Knee | Persona Without iASSIST Knee
Number analyzed (Participants) | 47 | 46
trays | 5.2 (2.2) | 4.9 (2.1)

7. Secondary Outcome: KSS - Objective Score at 6 Month Postoperatively
Description: KSS-Objective score is physician-derived component and allows for more than 100 points in patients with greater than 125° of flexion and a stable painless knee as outlined below. Lowest possible score is 0.
  Higher score means better outcomes.
Time Frame: 6 month postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Persona With iASSIST Knee | Persona Without iASSIST Knee
Number analyzed (Participants) | 42 | 41
score on a scale | 80.8 (13.9) | 77.2 (17.5)

8. Secondary Outcome: KSS-Patient Satisfaction at 6 Month Postoperatively
Description: KSS-Patient Satisfaction is patient-derived score and is a five-question 40-point scale that is collected preoperatively and at each follow-up visit. Lowest possible score is 0.
Time Frame: 6 month postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Persona With iASSIST Knee | Persona Without iASSIST Knee
Number analyzed (Participants) | 45 | 45
score on a scale | 24.6 (8.2) | 25.0 (8.3)

9. Secondary Outcome: KSS-function Score at 6 Month Postoperatively
Description: KSS-function score is patient-derived score and composed of four subgroups and has a maximum score of 100.
  "Walking and Standing" has a maximum value of 30 points, "Standard Activities" has a maximum of 30 points, "Advanced Activities" has a maximum of 25 points and "Discretionary Activities" has a maximum of 15 points.
  Lowest possible score is 0. Higher score means better outcomes.
Time Frame: 6 month postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Persona With iASSIST Knee | Persona Without iASSIST Knee
Number analyzed (Participants) | 42 | 41
score on a scale | 61.6 (23.7) | 61.5 (18.6)

10. Secondary Outcome: KSS-Patient Expectations at 6 Month Postoperatively
Description: KSS-Patient Expectations is patient-derived score and is a three-question fifteen-point scale that is collected pre-operatively and post-operatively. The pre-operative questions reflect the patient's opinion on the extent to which the patient expects that operation will improve knee pain, and ability to perform activities of daily living and recreational activities. The post-operative questions reflect the extent to which postoperative outcome has met the patient's pre-operative expectations with respect to pain and function.
  The score ranges from 3 to 15. Higher score means better outcomes.
Time Frame: 6 month postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Persona With iASSIST Knee | Persona Without iASSIST Knee
Number analyzed (Participants) | 42 | 41
score on a scale | 9.5 (3.1) | 10.1 (2.5)

11. Secondary Outcome: Oxford Knee Score at 6 Month Postoperatively
Description: Patient Reported Outcome specific for knee disease. Score range from 0 to 48. Higher score means better outcome.
Time Frame: 6 month postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Persona With iASSIST Knee | Persona Without iASSIST Knee
Number analyzed (Participants) | 42 | 41
score on a scale | 36.2 (9.2) | 37.7 (6.9)

12. Secondary Outcome: EQ-5D-3L at 6 Month Postoperatively
Description: EQ-5D is patient reported outcome measure to score patient's health related quality of life with minimum score of -0.111 and maximum score of 1.000.
  Higher score means better outcomes.
Time Frame: 6 month postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Persona With iASSIST Knee | Persona Without iASSIST Knee
Number analyzed (Participants) | 42 | 41
score on a scale | 0.8 (0.2) | 0.8 (0.2)

ADVERSE EVENTS:
Time Frame: Surgery to 6 month postoperative visit
Arm/Group | Persona With iASSIST Knee | Persona Without iASSIST Knee
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/42 | 1/41
Other Adverse Events (participants affected / at risk) | 0/42 | 1/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Persona With iASSIST Knee (N=42) | Persona Without iASSIST Knee (N=41)
Malignant Lymphoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Persona With iASSIST Knee (N=42) | Persona Without iASSIST Knee (N=41)
Postoperative Supracondylar Fracture of femur (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT03227692/Prot_SAP_000.pdf